CLINICAL TRIAL: NCT00298844
Title: Prevalence of Macrovascular Disease in Type 2 Diabetes Mellitus: Left Ventricular Diastolic Dysfunction, Myocardial Ischemia and Peripheral Vascular Insufficient
Brief Title: Prevalence of Macrovascular Disease in Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Other Study IDs: 021
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2007-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Macrovascular disease; Diastolic dysfunction; Intima media thickness; Single- photon emission computed tomography (SPECT)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The study aim is to establish a consecutive population of newly referred type 2 diabetes mellitus patients and among these to describe the degree of macrovascular disease by evaluating left ventricular systolic and diastolic function (echocardiography), myocardial perfusion (single-photon emission computed tomography (SPECT)), the peripheral vascular perfusion (strain gauge toe blood pressure measurements and a ultrasound scan of the a. carotis communis). Further, the degree of microvascular disease will be evaluated (glomerular filtration rate assessment, fundus photography and biotesiometry). Finally the cohort will be followed the next two years to assess the prognostic value of the above-mentioned parameters

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 20 years.
* Fasting C-peptide > 300 pmol/l.

Exclusion Criteria:

* Verified medical history of macrovascular disease (stroke, myocardiac infarct, coronary revascularisation or strain gauge toe blood pressure < 30 mmHg).
* Suspected short lifespan because of malignant disease or end-stage kidney disease.
* Pregnancy or planned pregnancy during the study period.
* Body weight > 150 kg.
* Physical or mental disability not enabling participation in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2006-01; Study Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mikael K. Poulsen, PhD student, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Pedersen L, Nybo M, Poulsen MK, Henriksen JE, Dahl J, Rasmussen LM. Plasma calprotectin and its association with cardiovascular disease manifestations, obesity and the metabolic syndrome in type 2 diabetes mellitus patients. BMC Cardiovasc Disord. 2014 Dec 19;14:196. doi: 10.1186/1471-2261-14-196. PMID 25527236
- [Derived] Poulsen MK, Dahl JS, Henriksen JE, Hey TM, Hoilund-Carlsen PF, Beck-Nielsen H, Moller JE. Left atrial volume index: relation to long-term clinical outcome in type 2 diabetes. J Am Coll Cardiol. 2013 Dec 24;62(25):2416-2421. doi: 10.1016/j.jacc.2013.08.1622. Epub 2013 Sep 24. PMID 24076532
- [Derived] Poulsen MK, Nybo M, Dahl J, Hosbond S, Poulsen TS, Johansen A, Hoilund-Carlsen PF, Beck-Nielsen H, Rasmussen LM, Henriksen JE. Plasma osteoprotegerin is related to carotid and peripheral arterial disease, but not to myocardial ischemia in type 2 diabetes mellitus. Cardiovasc Diabetol. 2011 Aug 12;10:76. doi: 10.1186/1475-2840-10-76. PMID 21838881
- [Derived] Poulsen MK, Henriksen JE, Vach W, Dahl J, Moller JE, Johansen A, Gerke O, Haghfelt T, Hoilund-Carlsen PF, Beck-Nielsen H. Identification of asymptomatic type 2 diabetes mellitus patients with a low, intermediate and high risk of ischaemic heart disease: is there an algorithm? Diabetologia. 2010 Apr;53(4):659-67. doi: 10.1007/s00125-009-1646-7. Epub 2010 Jan 14. PMID 20225395
- [Derived] Poulsen MK, Henriksen JE, Dahl J, Johansen A, Gerke O, Vach W, Haghfelt T, Hoilund-Carlsen PF, Beck-Nielsen H, Moller JE. Left ventricular diastolic function in type 2 diabetes mellitus: prevalence and association with myocardial and vascular disease. Circ Cardiovasc Imaging. 2010 Jan;3(1):24-31. doi: 10.1161/CIRCIMAGING.109.855510. Epub 2009 Oct 21. PMID 19846730
- [Derived] Poulsen MK, Henriksen JE, Dahl J, Johansen A, Moller JE, Gerke O, Vach W, Haghfelt T, Beck-Nielsen H, Hoilund-Carlsen PF. Myocardial ischemia, carotid, and peripheral arterial disease and their interrelationship in type 2 diabetes patients. J Nucl Cardiol. 2009 Nov-Dec;16(6):878-87. doi: 10.1007/s12350-009-9118-5. Epub 2009 Aug 14. PMID 19685102